CLINICAL TRIAL: NCT06918093
Title: A Comparative Evaluation of Different Histopathological Indices of Mucosal Healing in Ulcerative Colitis, and Their Correlation With Clinical Follow-up Data
Brief Title: A Comparative Evaluation of Different Histopathological Indices of Mucosal Healing in Ulcerative Colitis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Mahmoud Mohamed, Principal Investigator, Assiut University
Other Study IDs: UC STUDY
Record Dates: First submitted 2025-03-30; First posted 2025-04-09 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
* To evaluate the histological activity and the presence of specific histopathologic features at diagnosis in ulcerative colitis patients before and after receiving treatment using the three most widely- used histological scoring indices (Gobeos score , Robarts Histopathologic Index and Nancy Index )
* To compare the findings of the three histopathological indices with each other as a trial to select the best, reproducible, easily and consistently applied system that could be adopted in routine pathological evaluation. Moreover, an attempt to introduce a novel customized method of histopathological evaluation could be carried out.
* To correlate the clinical and endoscopic follow up data of patient on treatment with the histopathological evaluation. This will be done in order to evaluate the possible predictive effect of histopathological evaluation on the disease course and hence as a tool to drive possible modification of the therapeutic choices

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic inflammatory disease of idiopathic origin affecting the rectum and colon. Patients classically manifest with rectal bleeding, diarrhea, tenesmus, urgency, abdominal pain, weight loss, fever, and malaise. Pathologically, it is defined by a continuous mucosal inflammation of the rectum and a variable extent of the colon, without granulomas on mucosal biopsies. The course of UC is characterized by periods of remission and relapsing. In patients with extensive or severe inflammation, acute complications such as severe bleeding and toxic megacolon, which can lead to perforation, may occur. Patients newly diagnosed with UC have a 5-year risk of colectomy of 10-35%, and ultimately, persistent and extensive inflammatory activity increases the long-term risk of dysplasia and colorectal cancer.

While treatment of patients with UC is primarily aiming to achieve clinical remission (CR) and endoscopic remission (ER), there is now interest in targeting histological healing (HH) in addition to CR, as symptoms may not reliably correlate with histological activity. Moreover, ER is not always an accurate indicator of histological healing. Furthermore, histological changes tend to lag behind CR after treatment. Accordingly, histological remission may be considered as an independent predictor of clinical relapse better than endoscopic appearances.

The Selecting Therapeutic Targets in Inflammatory Bowel Disease (STRIDE) II committee introduced a treat-to-target approach and proposed that the therapeutic target in UC should include clinical and patient-reported outcome remission, alongside endoscopic remission, with Mayo endoscopic subscore of 0. Histologic remission is not a formal target of medical therapy, but it is considered an "adjunct to endoscopic remission to represent a deeper level of healing.

However, Various studies have elucidated that histologic remission serves as a distinct treatment objective from endoscopic remission, offering a superior prediction of clinical remission. In few studies, histological remission seems to correlate with long-term clinical remission, better clinical outcomes, and a lower risk of intestinal dysplasia, even though significant data are still lacking.

Currently, about 30 histologic scoring systems in UC have been described and used for quantitative assessment, but 3 have recently undergone scientific validation namely the Gobeos score (GS), Nancy Index (NI) and Robarts Histopathologic Index (RHI). For histologic measurements of disease activity to affect clinical decision making, pathologists should agree upon which standardized features to report and the definitions of these parameters.

GS evaluates all aspects of mucosal injury seen in UC including crypt architecture, lamina propria chronic inflammation, lamina propria eosinophils, lamina propria neutrophils, intraepithelial neutrophils, crypt destruction, and surface epithelial injury.

The RHI was developed based on several reproducible features included in the final index (lamina propria chronic inflammation, lamina propria neutrophils, neutrophils in the epithelium, and surface epithelial injury). Although the RHI was specifically designed to be responsive and reproducible, it requires assessment of 4 features to arrive at a calculated score, which may reduce its clinical usefulness.

The NI is a stepwise 5-item index that evaluates lamina propria chronic inflammation (defined as lymphocytes, plasma cells, and eosinophils), neutrophilic inflammation, and ulcers.

It is unclear which of these histologic scoring indices is most useful in clinical practice. In this context, it is important that pathologists to include important, reproducible histologic features in a pathology report that could be correlated better with clinical management. In addition, the development and validation of novel histologic scoring systems, better correlate with CR and ER, should be tried out.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >18 years diagnosed with ulcerative colitis based on standard clinical, endoscopic, and histological criteria

Exclusion Criteria:

* Patients lost to follow-up and those with insufficient data

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - The study will include 60 cases of patients diagnosed clinically and pathologically as ulcerative colitis and received therapeutic regimen at Department of Internal medicine ,Gastroenterology unit .- Biopsies of those patients will be reevaluated using the three histopathological indices; Gobeos score, Nancy Index and Robarts Histopathologic Index on hematoxylin and eosin stained slides
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
A Comparative Evaluation of Different Histopathological Indices of Mucosal Healing in Ulcerative Colitis, and their Correlation with Clinical Follow-up Data | 4 months
  -- To correlate the clinical and endoscopic follow up data of patient on treatment with the histopathological evaluation. This will be done in order to evaluate the possible predictive effect of histopathological evaluation on the disease course and hence as a tool to drive possible modification of the therapeutic choices

CONTACTS AND LOCATIONS:
Overall Officials: Thanaa Sotouhy, Professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marchal-Bressenot A, Salleron J, Boulagnon-Rombi C, Bastien C, Cahn V, Cadiot G, Diebold MD, Danese S, Reinisch W, Schreiber S, Travis S, Peyrin-Biroulet L. Development and validation of the Nancy histological index for UC. Gut. 2017 Jan;66(1):43-49. doi: 10.1136/gutjnl-2015-310187. Epub 2015 Oct 13. PMID 26464414
- [Background] Jauregui-Amezaga A, Geerits A, Das Y, Lemmens B, Sagaert X, Bessissow T, Lobaton T, Ferrante M, Van Assche G, Bisschops R, Geboes K, De Hertogh G, Vermeire S. A Simplified Geboes Score for Ulcerative Colitis. J Crohns Colitis. 2017 Mar 1;11(3):305-313. doi: 10.1093/ecco-jcc/jjw154. PMID 27571771
- [Background] Peyrin-Biroulet L, Arenson E, Rubin DT, Siegel CA, Lee S, Stephen Laroux F, Zhou W, Finney-Hayward T, Sanchez Gonzalez Y, Shields AL. A Comparative Evaluation of the Measurement Properties of Three Histological Indices of Mucosal Healing in Ulcerative Colitis: Geboes Score, Robarts Histopathology Index and Nancy Index. J Crohns Colitis. 2023 Nov 24;17(11):1733-1743. doi: 10.1093/ecco-jcc/jjad087. PMID 37225135
- [Background] Le Berre C, Honap S, Peyrin-Biroulet L. Ulcerative colitis. Lancet. 2023 Aug 12;402(10401):571-584. doi: 10.1016/S0140-6736(23)00966-2. PMID 37573077
- [Background] Magro F, Estevinho MM, Valois A. Managing Ulcerative Colitis and Crohn's Disease: Should the Target Be Endoscopy, Histology, or Both? J Can Assoc Gastroenterol. 2023 Sep 23;7(1):46-58. doi: 10.1093/jcag/gwad034. eCollection 2024 Feb. PMID 38314174
- [Background] Pai RK, Khanna R, D'Haens GR, Sandborn WJ, Jeyarajah J, Feagan BG, Vande Casteele N, Jairath V. Definitions of response and remission for the Robarts Histopathology Index. Gut. 2019 Nov;68(11):2101-2102. doi: 10.1136/gutjnl-2018-317547. Epub 2018 Oct 26. No abstract available. PMID 30366909
- [Background] Shehab M, Al Akram S, Hassan A, Alrashed F, Jairath V, Bessissow T. Histological Disease Activity as Predictor of Clinical Relapse, Hospitalization, and Surgery in Inflammatory Bowel Disease: Systematic Review and Meta-Analysis. Inflamm Bowel Dis. 2024 Apr 3;30(4):563-572. doi: 10.1093/ibd/izad119. PMID 37541185
- [Background] Turner D, Ricciuto A, Lewis A, D'Amico F, Dhaliwal J, Griffiths AM, Bettenworth D, Sandborn WJ, Sands BE, Reinisch W, Scholmerich J, Bemelman W, Danese S, Mary JY, Rubin D, Colombel JF, Peyrin-Biroulet L, Dotan I, Abreu MT, Dignass A; International Organization for the Study of IBD. STRIDE-II: An Update on the Selecting Therapeutic Targets in Inflammatory Bowel Disease (STRIDE) Initiative of the International Organization for the Study of IBD (IOIBD): Determining Therapeutic Goals for Treat-to-Target strategies in IBD. Gastroenterology. 2021 Apr;160(5):1570-1583. doi: 10.1053/j.gastro.2020.12.031. Epub 2021 Feb 19. PMID 33359090